CLINICAL TRIAL: NCT07369232
Title: Cerebral Hemodynamic Effects of Oxygen and Antioxidants
Brief Title: Cerebral Hemodynamic Effects of Oxygen and Antioxidants (CHEOXANT)
Acronym: CHEOXANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: National Research Council Italy - Institute of Clinical Physiology (CNR-IFC) (Unknown); FBM Lab Konsult AB - Sweden (Unknown)
Responsible Party: Principal Investigator, Fabio Taccone, Head of Department of Intensive Care, Erasme University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CEP2024/460
Record Dates: First submitted 2025-09-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Oxygen; Hyperoxemia; Antioxidant; Cerebral Autoregulation; Oxidative Stress
Keywords: oxygen; antioxidant; vitamin c; ascorbic acid; hyperoxia; hyperoxemia; physiology; microcirculation; microperfusion; trancranial doppler; microparticles; cerebral autoregulation
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, single-blind, placebo-controlled, crossover physiological study. Each volunteer undergoes two sessions, spaced at least one week apart, receiving vitamin C in one session and a placebo in the other, in randomized order.
Who Masked: Participant
Masking Description: Participants are blinded to the intervention (placebo vs. vitamin C infusion). Investigators and care providers are not blinded due to the nature of the procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Pre-Treatment + Oxygen (Placebo Comparator): Participants receive an intravenous infusion of 250 mL saline (placebo) over 20 minutes, 30-60 minutes before breathing 100% oxygen for 30 minutes through a reservoir mask. Measurements are performed at baseline, immediately after oxygen, and 1 hour later (cerebral blood flow by transcranial Doppler and skin microperfusion, blood pressure, arterial blood gases, oxidative stress markers, and microparticles).
  Interventions: Other: Oxygen
- Vitamin C Pre-Treatment + Oxygen (Experimental): Participants receive an intravenous infusion of 2 g ascorbic acid (vitamin C - ascorbic acid) diluted in 250 mL saline over 20 minutes, 30-60 minutes before breathing 100% oxygen for 30 minutes through a reservoir mask. Measurements are performed at baseline, immediately after oxygen, and 1 hour later (cerebral blood flow by transcranial Doppler and skin perfusion, blood pressure, arterial blood gases, oxidative stress markers, and microparticles).
  Interventions: Other: Oxygen; Drug: Vitamin C (Ascorbic Acid)

INTERVENTIONS:
Other: Oxygen — 30 minutes of normobaric 100% oxygen via reservoir mask 15L/min
Drug: Vitamin C (Ascorbic Acid) — 2 g ascorbic acid (vitamin C - ascorbic acid) diluted in 250 mL saline over 20 minutes, 30-60 minutes before breathing 100% oxygen
  Arms: Vitamin C Pre-Treatment + Oxygen

SUMMARY:
This study is called CHE-OX-ANT (Cerebral Hemodynamic Effects of Oxygen and Antioxidants). It is a single-center, academic research project led by the Department of Intensive Care at Erasme Hospital (Université Libre de Bruxelles).

The study focuses on understanding how the brain and blood vessels react when a person breathes pure oxygen and how these effects may be influenced by giving vitamin C, an antioxidant. Oxygen is one of the most common treatments in hospitals. While it can be life-saving, too much oxygen may sometimes cause harmful effects, such as oxidative stress (an imbalance between damaging molecules called free radicals and the body's defenses). Antioxidants like vitamin C may help counteract these effects.

The goal of the study is to examine how a short period of high oxygen (30 minutes of 100% oxygen through a mask) affects cerebral hemodynamics, microcirculation, microperfusion, blood markers (levels of oxidative stress, antioxidant activity, and microparticles).

The study will also test whether giving vitamin C beforehand changes these responses compared to a placebo (saline solution).

Each volunteer will participate in two sessions, one week apart. Before each session, participants will receive either vitamin C (given intravenously) or a placebo (saline). They will not know which one they receive.

Then, they will breathe 100% oxygen for 30 minutes through a facial mask. Measurements will be taken at three times: before oxygen (t0), just after oxygen (t1), and 1 hour later (t2). These include: ultrasound of the brain's blood flow (transcranial Doppler), measurements of skin perfusion and blood samplings.

DETAILED DESCRIPTION:
Oxygen therapy is widely used in hospitals and critical care, but excessive oxygen levels (hyperoxemia) can have both beneficial and harmful effects. In the brain, high oxygen may improve oxygen delivery, but it can also trigger oxidative stress, inflammation, and vascular dysfunction, potentially worsening outcomes. Antioxidants, such as vitamin C (ascorbic acid), may counteract these harmful effects by neutralizing reactive oxygen species and restoring redox balance. The CHE-OX-ANT study aims to investigate the physiological effects of a short normobaric hyperoxic stimulus (30 minutes of 100% oxygen breathing) in healthy volunteers, with and without prior antioxidant administration. The primary focus is on oxidative stress markers and microparticle production, while secondary objectives include effects on cerebral blood flow, sublingual microcirculation, and skin perfusion.

This is a prospective, interventional, single-center, randomized, single-blind, placebo-controlled physiological trial conducted at Erasme Hospital, Brussels. Each subject will serve as their own control, undergoing two study sessions one week apart. The study will recruit 10-15 healthy adult volunteers. Eligible participants must be >18 years old, in good health, with no cardiovascular, neurological, hematological, or immunological disease. Exclusion criteria include smoking, pregnancy, BMI >25, or contraindications to oxygen or vitamin

At each session, participants will receive one of two randomized pre-treatments, administered intravenously 30-60 minutes before oxygen exposure:

Vitamin C group: 1-3 g ascorbic acid in 500 mL saline infused over 20 minutes. Placebo group: 500 mL of saline infused over 20 minutes. Following this, participants will breathe 100% oxygen for 30 minutes through a reservoir mask. Measurements will be obtained at three timepoints: baseline (t0), immediately after oxygen (t1), and 2 hours post-exposure (t2).

Cerebral hemodynamics: Transcranial Doppler ultrasonography. Skin perfusion: laser Doppler or infrared techniques. Blood samples: venous and arterial blood for oxidative stress, antioxidant status, microparticles, and arterial blood gas analysis.

Blood pressure: continuous invasive monitoring via a radial arterial catheter. Endpoints Primary endpoint: Change in oxidative stress and microparticle levels. Secondary endpoints: Changes in cerebral hemodynamics and skin perfusion. This exploratory study will provide new insights into how oxygen affects the brain and peripheral perfusion, and whether antioxidant administration modifies these effects. The results may contribute to optimizing oxygen therapy in critically ill patients, where oxygen is widely used but may sometimes cause harm.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Otherwise healthy, without known pathologies in the cardiovascular, neurological, immunological, renal hematological, or vascular systems.

Exclusion Criteria:

* Smokers
* Pregnant women
* BMI > 25
* Any reason to avoid vit. C
* Any reason to avoid breathing oxygen at high doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in circulating microparticle concentration (total MPs - EV) | t0 = baseline (before infusion/oxygen administration) t1 = immediately after 30 minutes of 100% O₂ t2 = 1 hour after the end of exposure (post-exposure)
  A composite extracellular vesicle (MPs - EV) outcome reflecting brain and cerebral endothelial responses to hyperoxia, quantified in plasma by flow cytometry. The composite index will be derived from the standardized (z-score) change from baseline of the following EV subpopulations:
  GFAP-positive EVs (astrocyte-derived EVs) Aquaporin-4 (AQP4)-positive EVs (astrocyte/BBB-related EVs) TMEM119-positive EVs (microglia-related EVs) VE-cadherin (CD144)-positive EVs (endothelial junction-related EVs) CD62E (E-selectin)-positive EVs (endothelial activation-related EVs) Each EV subpopulation will be quantified as concentration (EVs/µL plasma). For each participant and time point, individual EV concentrations will be normalized (z-transformed) and combined into a single composite EV score by averaging the standardized values.
  The reported metric will be the within-participant change in the composite EV score from baseline (Δt1-t0 and Δt2-t0).
Change in oxidative stress and antioxidant status | t0 = baseline (before infusion/oxygen administration) t1 = immediately after 30 minutes of 100% O₂ t2 = 1 hour after the end of exposure (post-exposure)
  A composite biochemical outcome reflecting systemic oxidative stress and antioxidant balance in response to hyperoxia and vitamin C administration. The composite index will be derived from the standardized (z-score) change from baseline of the concentrations of the erythrocyte biomarker of antioxidant defense in mg/dL.
  For each participant and time point, biomarker values will be normalized (z-transformed) and combined

SECONDARY OUTCOMES:
Change in cerebral hemodynamics and autoregulation composite index | t0 = baseline (before infusion/oxygen administration) t1 = immediately after 30 minutes of 100% O₂ t2 = 1 hour after the end of exposure (post-exposure)
  A composite outcome summarizing cerebral hemodynamic and autoregulatory responses to hyperoxia, derived from transcranial Doppler (TCD) and arterial blood pressure signals. Dynamic cerebral autoregulation index (Mx, unitless) calculated using a predefined MATLAB/Python algorithm.
  For each participant and time point, it will be expressed as change from baseline and standardized (z-score), then combined into a single composite score by averaging the standardized component changes. The reported metric will be the within-participant change in the composite index from baseline
Change in skin perfusion | t0 = baseline (before infusion/oxygen administration) t1 = immediately after 30 minutes of 100% O₂ t2 = 1 hour after the end of exposure (post-exposure)
  Skin microcirculation will be assessed at a standardized site (fingertip) under controlled ambient temperature and resting conditions. The primary and only reported variable will be skin microvascular blood flow, expressed in perfusion units (PU) and measured using a validated microcirculatory technique.
  For each participant and time point, values will be averaged over predefined short acquisition windows to reduce signal variability. The reported metric will be the within-participant change in skin perfusion from baseline, expressed as absolute change in PU (Δt1-t0 and Δt2-t0).
  Skin temperature and relative (%) changes will be monitored only for quality control purposes and will not be reported as outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Intensive Care - Erasmus Hospital - ULB, Anderlecht, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
At present, there is no confirmed plan to share individual participant data (IPD). If sharing is pursued, it would involve de-identified datasets limited to physiological parameters, oxidative stress markers, microparticle levels, and circulatory measurements. No personally identifiable information will be shared.